CLINICAL TRIAL: NCT05408078
Title: Become Your Own SLEEPexpert: a Behavioral Treatment Program for Insomnia in Patients With Psychiatric Disorders
Acronym: SLEEPexpert
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Principal Investigator, Christoph Nissen, Professor, University of Bern
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-01897
Record Dates: First submitted 2021-10-28; First posted 2022-06-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This project is a prospective randomized controlled clinical pilot trial with a cluster-crossover design involving two groups: An interventional group (TAU, plus SLEEPexpert) and a control group (TAU plus sleep monitoring).
Who Masked: Outcomes Assessor
Masking Description: Study participants and care providers cannot be blinded because they will notice whether they receive / deliver an actual treatment or a monitoring control. Due to the crossover cluster design (randomization of wards to either TAU plus sleep monitoring or TAU plus SLEEPexpert), patients who are on the same ward at the same time will not get in contact with patients who are in the other arm. Thus, contamination due to exchange between patients will be reduced as far as possible.
  Outcome assessors (interviewers) and data analysts will be blinded. In the respective documents and database entries, patients will be identified with a code. The key for assigning the codes to patients will not be known to the interviewers and data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - Treatment as Usual (TAU) + SLEEPexpert (Experimental): SLEEPexpert is a behavioral programme for insomnia.
  The TAU + SLEEPexpert group will receive a specific treatment for insomnia. This treatment will consist of the following three phases:
  1. a face-to-face treatment initiation (kick-off) guided by a medical doctor/ psychologist in a group format
  2. self-managed implementation of behavioral changes supported by the nursing team (individual brief contact during the week)
  3. self-management by the patients, potentially assisted by the Webapplication after discharge from the hospital.
  Interventions: Device: SLEEPexpert
- Control group - TAU + sleep monitoring (Other): In addition to TAU, patients in the control group (TAU + sleep monitoring) receive a smartphone app (sleep monitoring). No further interventions will be provided through this app.
  TAU comprises standard clinical care, including intensive daily contacts with health care providers on the wards, medical treatment, pharmacotherapy, psychotherapy in individual and group setting, nurse support, additional therapies such as music or ergotherapy and social support, informed by current guidelines for the respective disorder and adapted to individual needs. Of note, no change to any aspects of TAU will be made. Sleep monitoring will consist of daily sleep diary entries with the help of a smartphone app.
  Interventions: Other: TAU plus sleep monitoring

INTERVENTIONS:
Device: SLEEPexpert — SLEEPexpert 1.0 is the first version of an online Program to treat Insomnia. The internet-based self-help platform used for the implementation of CBT-I in this study has been developed by the University of Bern (Prof. Dr. Thomas Berger), has been used successfully in previous trials and has received a CE mark in 2018.
  The device is intended for patients with mental disorders and insomnia who are treated for mental disorders in a hospital or an outpatient unit. No specific training is needed to operate the application.
  There is no available clinical research data to date on exactly this product. However, the therapeutic content that is used in this study is based on Cognitive Behavioral Therapy for insomnia (CBT-I). This intervention has been found to be highly effective and without lasting adverse effects in many studies and is recommended for the treatment of insomnia in current clinical guidelines.
  Arms: Intervention group - Treatment as Usual (TAU) + SLEEPexpert
Other: TAU plus sleep monitoring — Treatment aus Usual and a Sleep Monitoring App will be used. This is already described in the Arm Section
  Arms: Control group - TAU + sleep monitoring

SUMMARY:
Comorbid insomnia represents a frequent health problem in patients with severe mental disorders, and cognitive behavioral therapy for insomnia (CBT-I) has been identified as the first line treatment. However, CBT-I has not sufficiently been implemented in acute psychiatry settings. Rather, patients are often overtreated with benzodiazepines or benzodiazepine receptor agonists, related to adverse effects and the risk of tolerance and dependency. This work aims to empower patients with severe mental disorders to take care of their own sleep health based on a pragmatic behavioral treatment program ("Become your own SLEEPexpert"). Implementation research strategies in collaboration with patients and health care providers were used to adaptat CBT-I components to the needs of psychiatric inpatients. Evidence for feasibility in an acute hospital setting and preliminary evidence for efficacy has been shown. ln the proposed project, the investigators aim to compare treatment as usual (TAU) + SLEEPexpert to TAU + sleep monitoring in a pilot randomized controlled trial. The objective is to target sleep to improve mental health and to investigate the efficacy of the SLEEPexpert programme for the improvement of sleep and mental health. Given the high burden of comorbid insomnia in psychiatry, the investigators believe that the presented work is of interest to basic scientists and clinicians and, potentially, of heightened public health relevance.

DETAILED DESCRIPTION:
- Standard operating procedures: patient recruitment

During the enrolment phase, all patients admitted to the participating wards of the UPD Bern will be screened in person. The screening will consist of a few questions regarding sleep, implemented into the routine clinical interview at enrolment, and filling in the insomnia severity index. Eligible patients will be contacted by study staff, informed about the study, and invited to participate. For further information about the study, a flyer containing the most important details will be given to the participants. The screening and enrolment process will be standardized across the wards to minimize the risk of selection bias.

- Standard operating procedures: data collection & data management Source data verification Quality assurance: data validation & registry procedures

Data is recorded and collected in paper CRFs as source documents. ECRFs will be given as an option for direct anonymized data entry from participants if feasible. The eCRFs will be created and stored on the database RedCap which is a database recommended by the Clinical Trial Unit Bern. Data entry from the source paper CRFs to eCRFs should only be performed by authorized personnel and data should be consistent with the available source documents. When this is not the case, a detailed explanation of the discrepancies should be provided. The principal investigator should ensure the accuracy, completeness, and timeliness of the data reported and sign off the completed eCRFs. In order to reflect the current patient status throughout the study, eCRFs will be kept up to date. This means that eCRFs should be completed no later than two weeks after a participant's visit and that data entry not should be delayed unnecessarily.

- Data checks

Data edit checks will be implemented into the EDC (electronic data capture) system (RedCap), limiting entries to appropriate, realistic values (e.g. not allowing future dates, missing values etc.). Furthermore, selected data points are cross-checked for plausibility with previously entered data for each individual participant. Before database lock, each PI will validate the collected data from his site with his signature.

- Quality assurance: Site monitoring & auditing

On-site monitoring will be part of the quality control activities implemented for this study. For the purposes of monitoring, the PI at the site will provide the monitor with access to study documentation, patient records, facilities and any other resources necessary. No site audits by the sponsor are planned for this study, but the sponsor reserves the right to perform such an audit should it be considered necessary.

- Standard operating procedures: reporting of adverse events

AEs will be categorized concerning the type of the reaction, severity, relatedness to the intervention, action taken, and outcome. Adverse events will be asked at every study timepoint.

The frequency of occurrence of adverse events of different categories will be analysed using descriptive statistics and compared between the two groups using Chi square tests.

The sponsor investigator will report to the Ethics Committee via BASEC device deficiencies that could have led to serious adverse events if suitable action had not been taken, intervention had not been made, or circumstances had been less fortunate within 7 days

Sample size assessment A power analysis was conducted with G-Power. Assuming an alpha error level of 0.05 (two-sided) and a power of 0.8, a total sample size of n=60 will be sufficient to detect a medium effect (Cohen's d=0.65). This is a pilot trial with the primary aim of collecting qualitative experience and preliminary efficacy data. A large confirmatory trial will be conducted if the results of this pilot trial are encouraging.

Plan for missing data If a patient withdraws consent for further study participation, the data collected up to the time point of withdrawal will be included in the study and no further data will be collected. The data of withdrawn participants will not be anonymized but will remain coded after analysis of the data set. For participants who discontinue the study intervention but do not withdraw from participation in the study, study visits and data collection will continue in the same way as for non-withdrawn participants. Dropouts before start of treatment (i.e. non-starters) will be replaced by recruitment of new participants. Multiple imputation will be used in case data are not available for more than 5-10% of the sample.

- Standard operating procedures: Data analysis & statistical analysis plan Primary Analysis

The primary outcome, i.e. the four overall scores of the ISI of all follow-up time-points will be analyzed with a mixed effects linear model. The model will take into account the hierarchical structure of the data: multiple ISI scores per patient and clusters (cross-over). Because of the complexity of the data and the small number of clusters the investigators assume that they will not be able to introduce random effects for patients and clusters. However, the first approach will still be a linear mixed model with the following co-variables: fixed intervention effect (TAU plus SLEEPexpert versus TAU plus sleep monitoring), fixed baseline ISI score effect, random patient effect (multiple ISI scores during follow-up), random cluster effect. Depending on model fit, the investigators may need to simplify the model and modify the random effects. This model is pre-specified and the rationale for switching will be made explicit. The analysis will be made after all data has been collected by one of the principal investigators.

Secondary Analysis

Continuous outcomes (Brief Symptom Inventory, Beck Depression Inventory) will also be analyzed by a mixed effects linear model using the same procedure used to estimate the primary outcome. Binary outcome data will be analysed using mixed effect logistic regression with odds-ratio as the effect measure. The number of hospitalizations will be also analyzed by a mixed effects model.

Data dictionary The detailed data dictionary can be found in the study protocol in the document section.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented diagnosis of acute insomnia, i.e. insomnia criteria according to ICD-10 for at least 2 weeks
* Insomnia Severity Index (ISI) total score ≥ 8, equivalent to relevant insomnia
* Inpatient in one of the two participating psychiatric wards in the UPD Bern
* Ability to understand the aims and procedures of the study
* Willingness to participate and ability to provide written informed consent

Exclusion Criteria:

* Incabability of judgement
* Inability to participate in a low-threshold behavioral treatment program, e.g. due to severe cognitive impairment or high symptom severity precluding participation (e.g., severe catatonic symptoms, massive hallucinations, acute endangerment to self or others, involuntary commitment). Note that the named symptoms will lead to exclusion only if they lead to inability to give informed consent or an inability to participate in the program. Excluded patients will be re-assessed regularly and included if symptoms improve and participation is possible at a later point in time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | change from time point T0 (study start) to T1 ( week 1),T2(week2), T3 (week12), T4 (week26)
  The Insomnia Severity Index (ISI) is a valid, reliable and change-sensitive self-rating questionnaire that is widely used as an outcome measure in clinical trials in insomnia research (scores from 0 to 28 with higher values indicative for more severe insomnia).

SECONDARY OUTCOMES:
Change in Brief Symptom Inventory (BSI) 18-items | change from time point T0 (study start) to T2 (week 2) and T4 (week26)
  The investigators chose the Brief Symptom Inventory, 18 items (BSI) because it is an efficient measure of general mental health. In this study, patients will suffer from different mental disorders including but not limited to depression, psychosis, anxiety and substance abuse.). A general measure, beyond the severity of specific disorders, is thus needed to picture changes in general mental health (scores from 0 to 72 with higher values indicative of a higher symptom severity).

OTHER OUTCOMES:
Exploratory Outcome: Change in Beck Depression Inventory (BDI) | change from time point T0 (study start) to T2 (week 2) and T4 (week26)
  Measurement of the severity of depressive symptoms (scores from 0 to 63 with higher values indicative for more severe depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Nissen, Prof.Dr., Principal Investigator — University Hospital of Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis JG, Gehrman P, Espie CA, Riemann D, Perlis ML. Acute insomnia: current conceptualizations and future directions. Sleep Med Rev. 2012 Feb;16(1):5-14. doi: 10.1016/j.smrv.2011.02.002. Epub 2011 May 18. PMID 21596596
- [Background] Gagnon C, Belanger L, Ivers H, Morin CM. Validation of the Insomnia Severity Index in primary care. J Am Board Fam Med. 2013 Nov-Dec;26(6):701-10. doi: 10.3122/jabfm.2013.06.130064. PMID 24204066
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT05408078/Prot_SAP_000.pdf